CLINICAL TRIAL: NCT06369337
Title: Ultrasound Study of the Submentonian Musculature and Its Relationship in the Development of Dysphagia After Invasive Mechanical Ventilation: a Single-center Cohort Study
Brief Title: Ultrasound Study of the Submentonian Musculature and Its Relationship in Dysphagia
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Teresa Fernandez Pardo, Principal investigator, Universidad Europea de Madrid
Other Study IDs: 014-24
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Dysphagia, Oropharyngeal; Deglutition Disorders; Mechanical Ventilation Complication
Keywords: Dysphagia; Ultrasonography; Deglutition disorders; Diagnostic Imaging; Mechanical ventilation
MeSH Terms: conditions — Deglutition Disorders | interventions — Ultrasonography; Deglutition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group control: undeveloped dysphagia
  Interventions: Diagnostic Test: Ultrasound
- Group cohort: Developed dysphagia
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — The physical function variables will be analyzed through the Medical Research Council (MRC) and Functional Status Score (FSS), as well as swallowing function variables through the Volume-Viscosity Swallow (VVS-T) and Functional Oral Intake Scale scales. (FOIS) and Gugging Swallowing Screen (GUSS). The ecographic measurements will be made of the thickness and echogenicity of the submental and tonue muscles, as well as hyolaryngeal kinematics. These measurements will be performed 48 hours from the start of the orotracheal intubation episode, 7 days and 14 days of mechanical ventilation. To enable the correlation of clinical and ultrasound variables, one more independent measurement will be performed within the first 24 hours after authorization of oral tolerance in the patient.
  Other Names: Physical function; Swallowing function

SUMMARY:
Acquired dysphagia is one of the most frequent complications suffered by patients in intensive care units (ICU) after orotracheal extubation. Ultrasound has proven to be a useful method in the morphological and kinematic exploration of the main swallowing structures. AIM: to evaluate, through ultrasound procedures, the evolution of the morphology of the tongue and muscles of the floor of the mouth and the hyolaryngeal kinematics in patients intubated >48h and to correlate these measurements with the possible development of acquired dysphagia. The incidence of dysphagia and ICU acquired weakness (ICUAW) in subjects with >48h of intubation and the relative risk factors associated with baseline characteristics and clinical variables will be described. METHODOLOGY: Design: Single-center cohort study (Ramón y Cajal University Hospital). Participants: subjects >18 years old, admitted to an intensive care unit (ICU), with >48 hours of orotracheal intubation who meet eligibility criteria. Outcomes: the study of socio-demographic and clinical variables related to ICU admission will be included. The physical function variables will be analyzed through the Medical Research Council (MRC) and Functional Status Score (FSS), as well as swallowing function variables through the Volume-Viscosity Swallow (VVS-T) and Functional Oral Intake Scale scales. (FOIS) and Gugging Swallowing Screen (GUSS). Measurements will be made of the thickness and echogenicity of the submental and tongue muscles, as well as hyolaryngeal kinematics

ELIGIBILITY:
Inclusion Criteria:

* • Subjects >18 years old.

  * Having received an episode of orotracheal intubation for >48h

Exclusion Criteria:

* • Congenital or acquired conditions of the Central Nervous System (CNS) such as stroke, traumatic brain injury, Parkinson's, multiple sclerosis, amyotrophic lateral sclerosis (ALS) or any other condition that may bias the attribution of dysphagia to factors other than exclusively clinical ones.

  * Involvement of the cranial nerves or the Peripheral Nervous System (PNS) as well as diseases of the neuromuscular junction such as Myasthenia Gravis or any other condition that may bias the attribution of dysphagia to other factors that are not exclusively clinical.
  * Neck morphology incompatible with exploration through ultrasound procedures.
  * Secondary musculoskeletal injuries, including vertebral fractures, unstable extremity fractures or any condition that requires absolute bed rest as prescribed by a doctor.
  * Malignant tumor lesions or previous head and/or neck surgeries.
  * Medical-surgical history due to pathology of the larynx, oropharynx and/or esophagus.
  * Diagnosis of dysphagia or swallowing disorders prior to the intubation episode with IMV.
  * Patients unable to eat orally, at least partially.
  * Known prior cognitive impairment upon admission to the ICU.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to any of these units who have required IMV for a period greater than 48 hours who meet the eligibility criteria
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Thickness of the submental muscles | Baseline, 7 days, 14 days and 24 hours after authorization of oral tolerance in the patient.
  A measurement of the thickness of the digastric muscles will be performed, which will range from the upper to the lower fascial limit of the muscular belly, in its thickest territory and perpendicular to the superficial fascia of the mylohyoid muscle. The measurement of the thickness of the mylohyoid musculature will be carried out in two locations: (1) immediately below the measurement obtained for the left digastric muscle, between the limits of the superficial and deep fascia that surround it and (2) in its central raphe. The measurement of the thickness of the geniohyoid and genioglossus muscles will be carried out in their most central location, with a perpendicular line drawn from the raphe of the mylohyoid to the inferior fascia of the tongue. Finally, the thickness of the tongue will be made from the lower to the upper fascial edge, on the same line drawn for the genihyoid and Genioglossal muscles.
Hyolaryngeal displacement | 24 hours after authorization of oral tolerance in the patient.
  the convex probe will be used, placed longitudinally along the midline that follows the arrangement of the throat and the prominence of the thyroid cartilage. Two hyperechoic lines will be located, separated from each other, corresponding to the hyoid bone (cranial) and the most superior aspect of the ossification of the thyroid cartilage (caudal), which offer a posterior acoustic shadow artifact. 3 repetitions of a swallowing maneuver of a bolus of 3mL of water will be requested, with a rest interval of 1 to 2 minutes. These maneuvers will be recorded in video format for subsequent analysis with Image J Software (v 1.37; National Institutes of Health, Rockville, MD, USA). Each video will be analyzed frame by frame, selecting the most representative of the distances "a" (distance at rest) and "b" (maximum hyolaryngeal approximation). The result of this variable will be expressed in centimeters (cm) and % of approximation.

SECONDARY OUTCOMES:
Muscle strength | 24 hours after authorization of oral tolerance in the patient.
  Medical Research Council (MRC) Scale: this is a valid and reliable measure of the level of global muscle strength, widely used in the context of critically ill patients. It consists of 6 manual tests rated 0 (total absence of contraction) and 5 (preserved muscle capacity) applied bilaterally on different muscle groups of the upper and lower extremity, including: shoulder abduction, elbow flexion, wrist extension, flexion hip, knee extension and ankle dorsiflexion.
Functional Status | 24 hours after authorization of oral tolerance in the patient.
  Functional Status Score for the ICU Scale (FSS-UCI): allows the evaluation of 5 basic functional tasks both in the critically ill patient and in the patient admitted to the ward and after being discharged from the hospital, which include: turning, transfer from supine to sitting, sitting at the edge of the bed, transferring from sitting to standing and walking.
  The minimum value is 0 (non functional) and the maximum value is 7 (very functional)
Swallowing function | 24 hours after authorization of oral tolerance in the patient.
  Volume-Viscosity Swallow Test Scale (VVS-T): The VVS-T scale is a valid and reliable method for the detection of dysphagia, consisting of a protocol designed to maintain the safety and effectiveness of the patient's swallowing and directing the detection of silent bronchial aspiration episodes. Evaluates 3 types of texture with different viscosity (liquid texture -water-, nectar and pudding) at 3 volumes (5mL, 10mL and 20mL) to detect signs associated with safety (tone of voice, cough or desaturation) and with the effectiveness of swallowing (lip seal, oral residue, fractional swallow or pharyngeal residue).
Swallowing function | 24 hours after authorization of oral tolerance in the patient.
  Functional Oral Intake Scale (FOIS): the FOIS scale is currently one of the clinical tools for the evaluation of swallowing most accepted by scientific literature. It offers 7 levels of functionality (minimum value is 0 (non functional and maxim value is 7, very functional) in decreasing order of severity, divided into several blocks depending on the type of feeding (oral exclusively or dependent on alternative feeding).
Swallowing function | 24 hours after authorization of oral tolerance in the patient.
  Gugging Swallowing Screen Scale (GUSS): the GUSS scale provides another valid and reliable clinical alternative for the assessment of dysphagia. This scale is divided into two parts, an indirect swallowing test (up to 5 points) and another direct swallowing test, in turn subdivided into 3 sections (up to 5 points each). The indirect swallowing test includes a vigilance phase, a cough/throat-clearing maneuver, and saliva swallowing. The direct swallow test specifically evaluates swallowing, involuntary coughing, drooling, and/or voice change during the ingestion of semisolids, liquids, and solids.
  In this scale the minimun value is 0 and the maximum value is 20.This test allows screening the severity of dysphagia as mild or absent with minimal risk of aspiration (20 points), mild with low risk of aspiration (15-19), moderate with risk of aspiration (10-14) and severe with high risk. suction (0-9).